CLINICAL TRIAL: NCT03884387
Title: The Use of a Decision Aid in the Choice of Surgery for Herniated Disc
Brief Title: The Use of a Patient Decision Aid in the Choice of Surgery for Herniated Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Stina Lykke Brogård Andersen, Ph.d. student, Spine Centre of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16/1586
Record Dates: First submitted 2019-01-03; First posted 2019-03-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Herniated Disk
Keywords: Shared Decision Making, Lumbar Herniated Disk
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of a Patient Decision Aid (Experimental): A Patient Decision Aid is used in this arm in the clinical encounter. A tool designed to facilitate shared decision making when patients choose between surgical and non-surgical treatment for lumbar disc herniation .
  Interventions: Other: Patient Decision Aid
- Usual counceling (No Intervention): Usual counseling in the clinical encounter, when patients choose between surgical and non-surgical treatment for lumbar disc herniation .

INTERVENTIONS:
Other: Patient Decision Aid — The Patient Decision aid used in this project is a tool designed to facilitate shared decision making in patients with lumbar herniated disk. It is intended to complement counseling with health professionals and help patients become involved in decision making by making explicit the decision that needs to be made, providing information about the advantages and disadvantages of having or not having surgery, knowledge of treatment outcomes, and by clarifying personal values.
  Other Names: Beslutningshjælper©
  Arms: Use of a Patient Decision Aid

SUMMARY:
Even though surgery due to lumbar disc herniation (LDH) shows a more rapid relief of pain and recovery, the evidence of surgery being superior to conservative treatment in the long term is inconclusive. Involving patients in the decisions whether or not to have surgery is therefore essential. A small survey performed at our Spine Center however, showed that patients were often not fully involved in this treatment decision. Not being involved might lead patients to decision regret and unnecessary conflicts in the decision-making process. The purpose of this project is therefore to assess the effect of a newly developed patient decision aid (PtDA) to facilitate shared decision making (SDM), when patients choose between surgical or non-surgical treatment for LDH, on SDM, decisional conflict, decision regret and treatment outcomes in a randomized controlled trial. The project is performed at Center of Spine Surgery & Research, Middelfart. Inclusion and one month follow up is already completed and one year follow-up data currently being collected.

DETAILED DESCRIPTION:
Purpose of the project

The overall purpose of this study is to assess the effectiveness of a generic PtDA-template adapted to patients choosing between surgical and non-surgical treatment for LDH, on SDM, decisional conflict, decision regret and treatment outcomes in a randomized controlled trial. Development of an effective PtDA has the potential to decrease patients' decision regret and optimize treatment results and thereby in the future lead to higher patient satisfaction and fewer patient complaints. Using a generic PtDA-template, makes it feasible to adapt the used method to other spine-departments or other orthopedic-surgeries.

Background

Shared decision making (SDM) is a systematic approach aimed at improving patient involvement in preference-sensitive health care decisions. It is a process, wherein clinicians actively involve patients during the task of making decisions , based on best clinical evidence and patients' informed preferences.

Most people with lumbar disc herniation (LDH) improve with nonsurgical treatment. However, in Denmark, patients with ongoing severe pain and disability after 12 weeks of conservative care are recommended a surgical evaluation. Apart from the presence of a neurologic deficit, there are no clearly defined indications for surgery. A variety of factors, such as level of pain, walking capacity or functional limitations, can influence the judgment of the physician to advocate surgery or not. Indications for surgery are thus assessed, for each particular patient, by the individual surgeon. Even though surgical patients show a more rapid relief of pain and recovery, the evidence of surgery being superior to conservative treatment in the long term is nevertheless inconclusive. This underlines the concept that the choice of having surgical or non-surgical treatment for LHD is preference sensitive, meaning that treatment options should be offered and should matter to patients. A qualitative study by Andersen showed that the current lack of evidence for a superior treatment choice and the presence of uncertainties in risks and benefits are important to discuss with patients with LDH. Currently, there are no standard procedures used to actively involve patients in such decisions. SDM is required to accomplish the preference sensitive approach for patients with LDH.

Patient decision aids (PtDA) are tools designed to facilitate SDM, and are intended to complement counseling with health professionals. Such a tool could help patients become involved in decision making by making explicit the decision that needs to be made, providing information about the advantages and disadvantages of treatment options (or tests), knowledge of treatment outcomes, and by clarifying personal values. Decision Aids compared to usual care seems to improve decision quality and patient knowledge regarding options and reduce their decisional conflict. Some studies also show that PtDAs enable patients to be more actively involved in decision making, and improve the accuracy of risk perceptions when probabilities are included A few English tools have already been designed for patients with LDH. However, these tools were designed to prepare the patients, prior to consultation with a physician and not, as intended in this project, to be used in the clinical encounter. Therefore, prior to this study a PtDAs have been designed and tested for use in spine surgery in a Danish context.

Study 1 - Does the use of a decision aid in a spine surgery clinic facilitate SDM?

Objectives

The Objectives are to determine whether the use of a DA is superior to standard consultation, in terms of:

1. Involving and informing the patients in the decision of treatment.
2. Minimizing uncertainty, and other conflicting factors, when choosing treatment for herniated disc.

Methods

Design The study will be performed as a randomized controlled trial (RCT). Ten surgeons will be allocated to either using or not using a DA in the surgery clinic, in a 1:1 ratio.

Intervention The intervention is the use of a PtDA for LDH, in a routine doctor-patient consultation, by a trained spine surgeon. All surgeons randomized to use the PtDA will go through a training session held by educators in communication, who is specialized in SDM.

Study population Study subjects will be recruited from Center for Spine Surgery and Research, Lillebaelt Hospital, Middelfart, amongst patients being a candidate for primary discectomy for a LDH from L1-S1.

Data will be collected post consultation in both arms, as the patients exit the consultation.

Statistics (see study 2)

Study 2 - Does the use of a decision aid in a spine surgery clinic improve outcomes?

Objectives

The objectives are to determine if there is a correlation between the use of a DA in the consultation and:

1. Better recovery after treatment, measured by leg pain (VAS leg), back pain (VAS back), ODI and EQ5D, one month and one year after spine surgery.
2. The level of decisional regret one month and one year after chosen treatment.

Methods

Design, intervention and study-population will be the same as in study 2. However, if patients end up with other surgery than discectomy they will be excluded from the study.

Statistical analysis

As the DQW-HD, DCS, ODI, EQ-5D and VAS Leg and Back pain scores are long ordinal scales, differences in scores, between the groups will be tested using nonparametric Mann-Whitney test for independent samples. Sample size rationale was powered from the main outcome variable in study 3 VAS-leg. Allowing for 30% dropout before completing the study, we need to enroll 70 patients in each arm. All Statistical analyses will be performed using Stata v. 14.0.

Research plan The inclusion started in May 2017. All the patients in the RCT are included and one month follow-up data are collected. Collection of one year follow-up data will has also begun.

Practical framework

All Spine surgeons at the surgery department accepted to participate in the study. Patients were recruited by these surgeons. The research department assists with data-collection at one month and one year follow-up.

Publication and dissemination of results

Results will be published in national and international peer-reviewed journals (i.e. The Spine, The Patient - Patient-Centered Outcomes Research) and presented at national and international conferences (i.e. Dansk Ortopædkirurgisk Selskabs årsmøde (DOS), International Shared Decision Making conference (ISDM), International Conference on Communication in Health Care (ICCH).

Ethical aspects

The study will be conducted according to Danish ethical principles, and notified at the Danish Data Protection Agency. Participants will be given written information about the purpose of the study and will sign an informed consent before the first questionnaires are completed. Surgeons give oral consent. Apart from the use of a PtDA in the consultation, all patients in the study receive "usual care". No changes are made in relation to which clinicians the patients meet or offered treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by a surgeon in the Center for spine surgery and research, SLB.
* Clinical symptoms and concordant MRI findings of a LDH from L1 to S1 with possible indication for primary discectomy surgery, assessed by an experienced spinal surgeon
* Age >18
* Able to understand and read Danish
* Informed consent

Exclusion Criteria:

* General contra-indication for spine surgery
* Diagnosis of psychiatric disorder
* Manifest paresis disorder
* Previous spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Decision Quality worksheet -for herniated disc (DQW-HD v.2.0) | Meassured right after the surgeon-patient consultation
  Decision quality is defined as the extent to which treatments reflect the considered preferences of wellinformed patients and how well it is implemented. Decision quality worksheet - HD include decision-specific items to assess:
  1. knowledge, or the extent to which patients are informed
  2. patients' goals, concerns and preferred treatment. These items can then be used to calculate concordance, or the extent to which patients' receive treatments that match their goals.
  3. the decision making process, or the extent to which providers engage patients in decisions about their care.
  The three aspects are reported on separately, as a total knowledge score, a concordance (or in some cases dissonance) score, and a decisions process score.
  In this study only the knowledge and the process score is used. A total score is summed for each of the aspects ranging from 0-100 % with higher scores indicating a higher knowledge or a more shared decision- making process respectively.

SECONDARY OUTCOMES:
Decisional conflict scale | Meassured right after the surgeon-patient consultation
  The decisional conflict scale (DCS) measures personal perceptions of:
  1. uncertainty in choosing options;
  2. modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and
  3. effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
  A total score is presented ranging from 0-100 with 0 indicating no decisional conflict and 100 extremely high decisional conflict.
Visual Analog Scale (VAS) leg | One month and one year after decision is made
  The Visual Analogue Scale (VAS) consists of a straight line (10 cm of length) with the endpoints defining the limits 'no pain at all' to the left and 'pain as bad as it could be' to the right. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the patient's pain. A score is given ranging from 0-100 mm. A higher score indicates greater pain intensity.
Decisional Regret Scale | One month and one year after decision is made
  The Decision Regret Scale (a 5-item scale) measures "distress or remorse after a [health care] decision. A total score is presented ranging from 0-100 with 0 indicating no regret and 100 means high regret.
Oswestry Disability Index | One year after the decision is made
  This questionnaire has been designed to give information as to how patients back or leg pain is affecting their ability to manage in everyday life. The test is considered the 'gold standard' of low back functional outcome tools. A total score is presented ranging from 0-100 with 0 indicating no regret and 100 means high regret.
European Quality of life - 5 Dimensions (EQ-5D) | One year after decision is made
  EQ-5D is a standardized/generic measure of health status. It consists of 5 dimensions. Each of the dimensions are divided into 5 levels of perceived problems. A health state is defined by combining 1 level from each of the 5 dimensions. Each state is referred to in terms of a 5 digit code. In this study an idex value is found using the UK EQ-5D-5L index, which can define 3125 (=55) different health states. The value lies between -0.624 - 1.0, with higher index indicating better health state/quality of life and vice versa. (0.0 indicates death and -0,293 is beeing unconscious).

CONTACTS AND LOCATIONS:
Overall Officials: Stina B Andersen, MHS, Principal Investigator — Sygehus Lillebaelt
Locations (1):
- Middelfart spine surgery research department, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared with other researchers